CLINICAL TRIAL: NCT04359927
Title: Long-term Effects of Coronavirus 2019 Disease on the Cardiovascular System in Patients Who Have Undergone a Diagnostic Nasopharyngeal Swab for SARS-CoV-2. CV COVID-19 Registry
Brief Title: Long-term Effects of Coronavirus Disease 2019 on the Cardiovascular System: CV COVID-19 Registry
Acronym: CV-COVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Luis Ortega Paz, Principal Investigator, Hospital Clinic of Barcelona
Other Study IDs: HCB/2020/0457
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Sars-CoV2; Covid19; Cardiovascular Diseases; Cardiovascular Risk Factor
Keywords: Sars-CoV2; Covid19; Cardiovascular death; Cardiovascular Diseases; Cardiovascular Risk Factor
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-CoV2/Covid-19 (cases): Patients with detectable real-time reverse transcriptase-polymerase chain reaction for SARS-CoV2/Covid-19.
- No SARS-CoV2/Covid-19 (controls): Patients with undetectable real-time reverse transcriptase-polymerase chain reaction for SARS-CoV2/Covid-19.

SUMMARY:
Patients presenting with the coronavirus-2019 disease (COVID-19) have a very high risk of cardiovascular adverse events, including death from cardiovascular causes. Unfortunately, there are no reliable statistics on the frequency and severity of these complications during the index hospitalization. Moreover, the long-term cardiovascular outcomes of these patients are entirely unknown. The investigators aim to perform a registry of patients who have undergone a diagnostic nasopharyngeal swab for SARS-CoV-2 and determine their long-term cardiovascular outcomes.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is an infectious disease caused by severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) that has posed a significant threat to global health. Angiotensin-converting enzyme 2 (ACE2) has been identified as a functional receptor for coronaviruses, including SARS-CoV and SARS-CoV-2. SARS-CoV-2 infection is triggered by the binding of the virus spike protein to ACE2, which is highly expressed in the heart and lungs.

There are multiple connections between COVID-19 and the cardiovascular system. First, COVID-19 patients and pre-existing cardiovascular disease are at increased risk for serious adverse events. Second, the infection has been associated with multiple direct and indirect cardiovascular complications, such as acute myocardial injury, myocarditis, arrhythmias, and thromboembolism. Third, the therapies under investigation for COVID-19 may have cardiovascular side effects. There is clear scientific evidence linking COVID-19 with cardiac damage, with a subsequent impact on mortality from any cause. The reasons for increased mortality in patients with COVID-19 and heart damage are not fully understood.

The long-term prognosis for patients who have had COVID-19 is entirely unknown. Previous experience with SARS-CoV suggests that both the underlying disease and its treatment could be associated with a worse cardiovascular prognosis. In a study of 25 survivors of SARS-CoV, at 12 years of follow-up, altered lipid metabolism was found. Similarly, viral diseases such as influenza A are associated with increased cardiovascular mortality after infection.

For the reasons stated above, the investigators consider that patients who presented COVID-19 have a high risk of long-term cardiovascular adverse events such as cardiac death, myocardial infarction, stroke, heart failure, and cardiac arrhythmias. To test this hypothesis, the investigators aimed to perform a registry of patients who have undergone a diagnostic nasopharyngeal swab for SARS-CoV-2 and determine their long-term cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent a nasopharyngeal swab for real-time reverse transcriptase-polymerase chain reaction for SARS-CoV2 in the participating institutions will be included.
Sampling Method: Non-Probability Sample
Enrollment: 4538 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular mortality | 1-year
  Cardiovascular mortality is defined according to the Academic Research Consortium-2 and will be independently adjudicated by a Clinical Events Committee.

SECONDARY OUTCOMES:
Acute myocardial infarction | 1-year
  Acute myocardial infarction is defined according to the Academic Research Consortium-2.
Stroke | 1-year
  Stroke is defined according to the Academic Research Consortium-2.

OTHER OUTCOMES:
Heart failure hospitalization | 1-year
  Documented hospital admission due to heart failure
Pulmonary embolism | 1-year
  Documented by a chest computed tomography
Cardiac arrhythmias | 1-year
  Documented hospital admission due to any cardiac arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Luis Ortega Paz, MD, PhD, Principal Investigator — Hospital Clínic of Barcelona; Salvatore Brugaletta, MD, PhD, Study Director — Hospital Clínic of Barcelona; Manel Sabaté, MD, PhD, Study Chair — Hospital Clínic of Barcelona
Locations (1):
- Hospital Clínic of Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
Will be made available upon request.

REFERENCES:
- [Background] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Circulation. 2018 Jun 12;137(24):2635-2650. doi: 10.1161/CIRCULATIONAHA.117.029289. PMID 29891620
- [Background] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Background] Arevalos V, Ortega-Paz L, Fernandez-Rodriguez D, Alfonso Jimenez-Diaz V, Rius JB, Campo G, Rodriguez-Santamarta M, de Prado AP, Gomez-Menchero A, Diaz Fernandez JF, Scardino C, Gonzalo N, Pernigotti A, Alfonso F, Jesus Amat-Santos I, Silvestro A, Ielasi A, Maria de la Torre J, Bastidas G, Gomez-Lara J, Sabate M, Brugaletta S; CV COVID-19 Registry Investigators. Long-term effects of coronavirus disease 2019 on the cardiovascular system, CV COVID registry: A structured summary of a study protocol. PLoS One. 2021 Jul 29;16(7):e0255263. doi: 10.1371/journal.pone.0255263. eCollection 2021. PMID 34324524
- [Derived] Ortega-Paz L, Arevalos V, Fernandez-Rodriguez D, Jimenez-Diaz V, Baneras J, Campo G, Rodriguez-Santamarta M, Diaz JF, Scardino C, Gomez-Alvarez Z, Pernigotti A, Alfonso F, Amat-Santos IJ, Silvestro A, Rampa L, de la Torre Hernandez JM, Bastidas G, Gomez-Lara J, Bikdeli B, Garcia-Garcia HM, Angiolillo DJ, Rodes-Cabau J, Sabate M, Brugaletta S; CV COVID-19 registry investigators. One-year cardiovascular outcomes after coronavirus disease 2019: The cardiovascular COVID-19 registry. PLoS One. 2022 Dec 30;17(12):e0279333. doi: 10.1371/journal.pone.0279333. eCollection 2022. PMID 36583998